CLINICAL TRIAL: NCT06949475
Title: Comparison of Dual Task and Upper Extremity Performance in Children With Myelomeningocele and Typically Developing Peers
Brief Title: Dual Task and Upper Extremity Performance in Children With Myelomeningocele
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: AIBU-FTR-ST-04
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Meningomyelocele
Keywords: Meningomyelocele; Dual task; Upper extremity performance
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meningomyelocele Group: Individuals between the ages of 7-18 years with a diagnosis of meningomyelocele
  Interventions: Diagnostic Test: Single Task (Box and Block Test); Diagnostic Test: Single Task (Nine Hole Peg Test); Diagnostic Test: Dual Task (Box and Block Test-Kognitif Task); Diagnostic Test: Dual Task (Nine Hole Peg Test-Kognitif Task); Diagnostic Test: Dual Task (Box and Block Test-Motor Task); Diagnostic Test: Dual Task (Nine Hole Peg Test-Motor Task); Diagnostic Test: ABILHAND-Kids; Diagnostic Test: Functional Mobility Scale (FMS); Diagnostic Test: Myelomeningocele Functional Classification System (MMFC); Diagnostic Test: Modified Mini Mental Test (MMMT)
- Typical Developing Group: Typically developing individuals between the ages of 7-18, who do not have any musculoskeletal system problems and who volunteer to participate in the study, who do not have a chronic neurological, cardiovascular or orthopedic disease
  Interventions: Diagnostic Test: Single Task (Box and Block Test); Diagnostic Test: Single Task (Nine Hole Peg Test); Diagnostic Test: Dual Task (Box and Block Test-Kognitif Task); Diagnostic Test: Dual Task (Nine Hole Peg Test-Kognitif Task); Diagnostic Test: Dual Task (Box and Block Test-Motor Task); Diagnostic Test: Dual Task (Nine Hole Peg Test-Motor Task); Diagnostic Test: ABILHAND-Kids

INTERVENTIONS:
Diagnostic Test: Single Task (Box and Block Test) — The test requires a wooden box divided into two compartments and 150 blocks (2.5 cm tall). When administering the test, the evaluator should be aware of whether the child's fingertips move from one compartment to the other. The number of blocks passed from one side of the box to the other in one minute determines the level of the skill. It is done separately for right and left hand. The number of cubes thrown in 1 minute gives the score.
Diagnostic Test: Single Task (Nine Hole Peg Test) — The 9-hole peg test is a standardized test that measures fine dexterity against time. It is simple to administer and is a valid and reliable method of assessment. Both hands are tested in the assessment. The child is first asked to place 9 sticks of 3.2 cm in length into the holes on the platform as quickly as possible with the dominant hand and the time from the start command until the last stick is placed is recorded. Then, with the same hand, he/she is asked to pick up the sticks in order and the time to remove all the sticks is recorded in seconds. The same procedure is repeated with the other hand.
Diagnostic Test: Dual Task (Box and Block Test-Kognitif Task) — Box Block Test-for the cognitive task assessment, the individual will be asked to count animal names while performing the test.
Diagnostic Test: Dual Task (Nine Hole Peg Test-Kognitif Task) — 9 Hole Peg Test-for the cognitive task assessment, the individual will be asked to count backwards from 20 one by one while performing the test
Diagnostic Test: Dual Task (Box and Block Test-Motor Task) — For the Box Block Test-motor task assessment, the individual will be asked to keep a rhythm by tapping the table with the fingers on the other side while performing the test. The number of blocks passed from one side to the other side of the box divided into two in one minute will be determined and recorded.
Diagnostic Test: Dual Task (Nine Hole Peg Test-Motor Task) — 9 Hole Peg Test-for motor task assessment, the individual will be asked to bend and unbend the other elbow while performing the test.
Diagnostic Test: ABILHAND-Kids — The Abilhand Kids Hand-Related Ability Scale will be used to assess the use of upper extremities in Activities of Daily Living (ADL). The scale includes 21 sub-items. Sub-items are scored as 0; cannot do, 1; has difficulty in doing and 2; can easily do. The questions are usually answered by the parent, but can also be answered by the child if the child is old enough and cognitive level is appropriate.
Diagnostic Test: Functional Mobility Scale (FMS) — The child's walking ability is assessed at 3 different distances (5 meters (home), 50 meters (school), 500 meters (community)). The assessment at all three distances is graded on a scale of 1-6, with wheelchair mobilization 1 and independent ambulation 6. It is indicated as (C) if the distance can be covered by crawling and (N) if the distance cannot be covered by any other means. The assessment is done through an interview with the family. The child is not observed.
  Groups: Meningomyelocele Group
Diagnostic Test: Myelomeningocele Functional Classification System (MMFC) — The Myelomeningocele Functional Classification System (MMFC) is a 4-level system that classifies individuals with myelomeningocele according to their functional capacity. The functional status of children in Level 1 is more inadequate than in other levels. Functional status improves as the level increases.
  Groups: Meningomyelocele Group
Diagnostic Test: Modified Mini Mental Test (MMMT) — The Modified Mini Mental Test (MMMT) is used to screen for cognitive dysfunctions in children, to assess the severity of impairments and to determine changes over time. It has been reported that the test is a suitable tool for examining cognitive functions in children from the age of 4 and can be easily included in general neurological examinations of children. The test, which takes 5 to 10 minutes to administer, assesses 5 cognitive domains, including orientation, memory, concentration, language function and measures of structural ability. The total score in this test reaches a plateau at approximately 9-10 years of age. In children over 10 years of age, scores below 27 out of a total of 35 points are indicative of mental retardation.
  Groups: Meningomyelocele Group

SUMMARY:
Myelomeningocele is a neural tube defect caused by the failure of the neural tube to close in the caudal part. The exposed spinal cord in myelomeningocele usually causes neural damage. Children with myelomeningocele have varying degrees of disability depending on the level of lesion and the presence of CNS-related anomalies. Lower limb weakness, sensory loss or deformity, and impaired bowel and bladder function are common disabilities that need to be managed. Performing multiple tasks simultaneously is a necessity in the daily lives of both adults and children. Although the majority of children with myelomeningocele lack the ability to ambulate and spend most of the day sitting, they have to perform dual tasking while performing activities of daily living as in all children. In the literature, dual task performance has been evaluated in many studies in adult individuals with diseases such as Multiple sclerosis, Stroke, Parkinson's, etc. However, there are few studies in the pediatric population in the literature. Most of the studies conducted in children include children with cerebral palsy and there are almost no studies in children with myelomeningocele. Therefore, the aim of this study was to compare dual task and upper extremity performance in children with myelomeningocele to typically developing peers.

DETAILED DESCRIPTION:
Within the scope of the study, socio-demographic information of the individuals will be recorded first. Afterwards, the Box Block Test and 9-hole peg test will be performed for single task assessment. The children will be seated on a chair with back support and before the test starts, all the details about the application will be explained to the person and the person will be given the opportunity to make a trial and if there are mistakes, they will be warned and then the actual evaluation will be started.

After the single task evaluation, the dual task performance will be evaluated. When testing dual task performance, participants will be asked to perform both tasks without prioritizing them and to do their best. However, they will also be instructed not to pause for reflection. A rest interval of at least 3 minutes will be given between all tests. Dual task complexity of the given upper limb functions will be measured by calculating the 'dual task effect' for both tasks. The formula used to calculate the dual task effect is as follows: Dual Task Effect=(Dual Task-Single Task/Single Task)x 100. If the result is positive, it is assumed that there is an improvement in the dual task conditions; if it is negative, it is assumed that there is a decrease in the dual task conditions. The results of children's performance will be recorded in the relevant table in the demographic data form

ELIGIBILITY:
Inclusion Criteria:

For children with meningomyelocele

* To be between the ages of 7-18
* To have been diagnosed with meningomyelocele
* To have scored 27 points or more on the modified mini mental test

For children with typical developing

* Being between the ages of 7-18 years
* Having no typically developing musculoskeletal problems and volunteering to participate in the study
* Not having a chronic neurological, cardiovascular or orthopedic disease
* Having a score of 27 or above on the modified mini mental test

Exclusion Criteria:

For children with meningomyelocele

* Not agreeing to participate in the study,
* Having undergone surgery or Botolunium toxin administration within the last six months
* Having suffered a fracture of the upper extremity within the last six months

For children with typical developing

* Having severe visual or hearing impairment
* Having attention problems to the extent that they cannot understand the assessment instructions
* Having a musculoskeletal, cardiovascular, pulmonary, metabolic or other disease severe enough to prevent participation in the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with meningomyelocele and typically developing peers who agreed to participate in the study and met the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Dual Task (Box and Block Test-Motor Task) | through study completion, an average of 1 year
  The test requires a wooden box divided into two compartments and 150 blocks (2.5 cm tall). When administering the test, the evaluator should be aware of whether the child's fingertips move from one compartment to the other. The number of blocks passed from one side of the box to the other in one minute determines the level of the skill. It is done separately for right and left hand. The number of cubes thrown in 1 minute gives the score. For the Box Block Test-motor task assessment, the individual will be asked to keep a rhythm by tapping the table with the fingers on the other side while performing the test. The number of blocks passed from one side to the other side of the box divided into two in one minute will be determined and recorded.
Dual Task (Box and Block Test-Kognitif Task) | through study completion, an average of 1 year
  The test requires a wooden box divided into two compartments and 150 blocks (2.5 cm tall). When administering the test, the evaluator should be aware of whether the child's fingertips move from one compartment to the other. The number of blocks passed from one side of the box to the other in one minute determines the level of the skill. It is done separately for right and left hand. The number of cubes thrown in 1 minute gives the score. Box Block Test-for the cognitive task assessment, the individual will be asked to count animal names while performing the test.
Dual Task (Nine Hole Peg Test-Motor Task) | through study completion, an average of 1 year
  The Nine Hole Peg test is a standardized test that measures fine dexterity against time. It is simple to administer and is a valid and reliable method of assessment. Both hands are tested in the assessment. The child is first asked to place 9 sticks of 3.2 cm in length into the holes on the platform as quickly as possible with the dominant hand and the time from the start command until the last stick is placed is recorded. Then, with the same hand, he/she is asked to pick up the sticks in order and the time to remove all the sticks is recorded in seconds. The same procedure is repeated with the other hand. 9 Hole Peg Test-for motor task assessment, the individual will be asked to bend and unbend the other elbow while performing the test.
Dual Task (Nine Hole Peg Test-Kognitif Task) | through study completion, an average of 1 year
  The Nine Hole Peg test is a standardized test that measures fine dexterity against time. It is simple to administer and is a valid and reliable method of assessment. Both hands are tested in the assessment. The child is first asked to place 9 sticks of 3.2 cm in length into the holes on the platform as quickly as possible with the dominant hand and the time from the start command until the last stick is placed is recorded. Then, with the same hand, he/she is asked to pick up the sticks in order and the time to remove all the sticks is recorded in seconds. The same procedure is repeated with the other hand. 9 Hole Peg Test-for the cognitive task assessment, the individual will be asked to count backwards from 20 one by one while performing the test

SECONDARY OUTCOMES:
Single Task (Box and Block Test) | through study completion, an average of 1 year
  The test requires a wooden box divided into two compartments and 150 blocks (2.5 cm tall). When administering the test, the evaluator should be aware of whether the child's fingertips move from one compartment to the other. The number of blocks passed from one side of the box to the other in one minute determines the level of the skill. It is done separately for right and left hand. The number of cubes thrown in 1 minute gives the score.
Single Task (Nine Hole Peg Test) | through study completion, an average of 1 year
  The Nine Hole Peg test is a standardized test that measures fine dexterity against time. It is simple to administer and is a valid and reliable method of assessment. Both hands are tested in the assessment. The child is first asked to place 9 sticks of 3.2 cm in length into the holes on the platform as quickly as possible with the dominant hand and the time from the start command until the last stick is placed is recorded. Then, with the same hand, he/she is asked to pick up the sticks in order and the time to remove all the sticks is recorded in seconds. The same procedure is repeated with the other hand.
ABILHAND-Kids | through study completion, an average of 1 year
  The Abilhand Kids Hand-Related Ability Scale will be used to assess the use of upper extremities in Activities of Daily Living (ADL). The scale includes 21 sub-items. Sub-items are scored as 0; cannot do, 1; has difficulty in doing and 2; can easily do. The questions are usually answered by the parent, but can also be answered by the child if the child is old enough and cognitive level is appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Tezcan, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu abant Izzet Baysal University, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No